CLINICAL TRIAL: NCT05179135
Title: Effects of Different Modalities of Postprandial Exercise on Glycaemia and Metabolism During and in the 24 Hours After Exercise in People with Type 1 Diabetes
Brief Title: Effects of Postprandial Exercise on Glycaemia and Metabolism in People with Type 1 Diabetes
Acronym: PRANDEX-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B6702021000244
Record Dates: First submitted 2021-12-03; First posted 2022-01-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Control (Active Comparator): Standardized meal, without exercise
  Interventions: Other: Postprandial exercise of different modalities
- Low-intensity walking (Experimental)
  Interventions: Other: Postprandial exercise of different modalities
- Moderate-intensity cycling (MOD) (Experimental)
  Interventions: Other: Postprandial exercise of different modalities
- High-intensity interval exercise (HIIT) (Experimental)
  Interventions: Other: Postprandial exercise of different modalities
- Intermittent high-intensity exercise (IHE) (Experimental)
  Interventions: Other: Postprandial exercise of different modalities

INTERVENTIONS:
Other: Postprandial exercise of different modalities — Physical exercise performed 60 minutes after a standardized meal, of different modalities (4 different modalities will be examined, as described in the Arms)

SUMMARY:
A cornerstone in the management and treatment of people living with type 1 diabetes (T1D) is to engage in regular physical exercise for a variety of health and fitness reasons. Despite these well-established benefits, many people with T1D experience their challenging glycaemic condition as a high barrier to exercise. The challenge of managing glycaemia around exercise together with fear of hypoglycaemia (FOH) remain major barriers to exercise in T1D patients, meaning that many are discouraged from exercise. If people with T1D wish to engage in exercise in a safe manner, a certain level of pre-planning before exercise is required in terms of insulin dosing and target glucose concentration.

Numerous research projects have been performed in the morning where participants exercise in the fasted state, for logistical reasons, because of easier insulin management in fasting conditions and a lower risk of hypoglycaemia during or after the exercise bout. However, in reality, advanced planning of exercise is not always possible, and many patients may also wish to exercise after their meal.

Hence, it is important to take into account the impact of prandial state on blood glucose responses to exercise in patients with T1D. While evidence on the importance of timing of exercise and on the benefits of postprandial exercise for improving glucose control is available in patients with type 2 diabetes, less studies have been conducted in T1D despite this being of high clinical importance.

Therefore, more insight is needed into the glycaemic and metabolic effects of different postprandial exercise modalities aiming to reduce the risk of hypoglycaemia and improve glucose control, both during and after exercise. Postprandial exercise can be a useful strategy to improve glycaemic control but research in T1DM is very scarce, with only few studies that have been conducted and optimal exercise regimens remaining unknown.

Summarizing, prandial state is an important factor to take into account in exercise in people with T1D, with glycaemic responses that substantially vary between fasted or postprandial exercise. Performing exercise in the postprandial period is of high clinical relevance however there is a scarcity of research in this area. Therefore, more studies that examine the glycaemic and metabolic effects of different modalities of postprandial exercise in people with T1D are needed. All of this aiming to simplify exercise-associated countermeasures and improve (postprandial) glucose control, and thereby reduce barriers to PA in this population.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for ≥ 2 years and negative C-peptide (<100pmol/l)
* Male and female aged 18-65 years old
* HbA1c <9% (at least two values in a row in the past year), based on analysis from the central laboratory unit of Ghent University Hospital.
* Insulin treatment: multiple daily injections (MDI) or continuous subcutaneous insulin infusion (CSII): insulin pump alone without connection to sensor, or sensor-augmented pump (SAP) with or without stop at/before low; however no hybrid closed-loop systems will be included).
* Able to understand study instructions and to provide written informed consent.

Exclusion Criteria:

* Physical or psychological disease likely to interfere with the normal conduct of the study as judged by the investigator.
* Body mass index >= 35 kg/m2.
* Self-monitoring of blood glucose (SBMG) with finger prick
* CSII with a hybrid closed-loop insulin pump
* Taking any medication that affects heart rate.
* Current treatment with drugs known to interfere with metabolism, e.g. systemic corticosteroids, SGLT2 inhibitors, glucagon-like-peptide 1 (GLP-1) receptor agonists, or metformin.
* Hypoglycaemic unawareness (Gold score ≥4) or having experienced any episode of a severe hypoglycaemic event within the last 6 months (i.e. need of third-party assistance).
* Known coronary or cerebral artery disease, i.e. history of angina pectoris, myocardial infarction (MI), stroke or any cardiovascular procedure.
* Severe non-proliferative and unstable proliferative retinopathy, based on medical record.
* Severe diabetic peripheral neuropathy (DPN) or autonomic neuropathy, based on medical record.
* Uncontrolled hypertension (>180/100 mmHg).
* Pregnant or planning to become pregnant during the study period (females)
* Breastfeeding (females).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
Change in blood glucose during exercise | 30 minutes (i.e. during exercise)
  Change in BG during exercise, calculated based on the participants' BG at the start of exercise and the last value measured at the end of exercise. (If the exercise is stopped early because of hypoglycaemia, the last exercise glucose value will be used for analysis.)

SECONDARY OUTCOMES:
Mean blood glucose during exercise and in the 30 min period after exercise. | 180 minutes
Incremental area under the blood glucose curve (iAUC) during exercise and in the 30 min period after exercise. | 180 minutes
Peak postprandial blood glucose (peak BG) concentration. | 120 minutes
Mean interstitial glucose concentration during the overnight period (12:00 AM - 06:00 AM), and in the 24 hours following exercise. | 24 hours
Incremental area under the interstitial glucose curve during the overnight period (12:00 AM - 06:00 AM), and in the 24 hours following exercise. | 24 hours
Incidence of hypoglycaemia during exercise, in the 30 min period after exercise, up to the late postprandial period (240 minutes after the meal), in the overnight period (12:00 AM - 06:00 AM), and the 24 hours following exercise. | 24 hours
Mean plasma lactate concentration during exercise and in the recovery period after the exercise session. | 180 minutes
Mean plasma free fatty acids concentration during exercise and in the recovery period after the exercise session. | 180 minutes
Mean plasma triglycerides concentration during exercise and in the recovery period after the exercise session. | 180 minutes
Mean plasma insulin concentration during exercise and in the recovery period after the exercise session. | 180 minutes
Plasma insulin area under the curve during exercise and in the recovery period after the exercise session. | 180 minutes
Mean plasma glucagon concentration during exercise and in the recovery period after the exercise session. | 180 minutes
Plasma glucagon area under the curve during exercise and in the recovery period after the exercise session. | 180 minutes
Mean plasma adrenaline concentration during exercise and in the recovery period after the exercise session. | 180 minutes
Plasma adrenaline area under the curve during exercise and in the recovery period after the exercise session. | 180 minutes
Mean plasma noradrenaline concentration during exercise and in the recovery period after the exercise session. | 180 minutes
Plasma noradrenaline area under the curve during exercise and in the recovery period after the exercise session. | 180 minutes
Mean plasma cortisol concentration during exercise and in the recovery period after the exercise session. | 180 minutes
Plasma cortisol area under the curve during exercise and in the recovery period after the exercise session. | 180 minutes
Mean plasma growth hormone concentration during exercise and in the recovery period after the exercise session. | 180 minutes
Plasma growth hormone area under the curve during exercise and in the recovery period after the exercise session. | 180 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No